CLINICAL TRIAL: NCT05043454
Title: Improving Age-Related Cognitive Decline With Exercise in Hypertensive Older Adults: A Pilot Study to Investigate A Retinal Microvascular Biomarker and the Role of IGF
Brief Title: Improving Age-Related Cognitive Decline With Exercise in Hypertensive Older Adults
Acronym: DECLARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ronald M. Lazar, PhD, Professor of Neurology, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300007742
Record Dates: First submitted 2021-08-25; First posted 2021-09-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — High-Intensity Interval Training; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vascular Density Improvement in Hypertensive Participants (Experimental): Participants will undergo baseline visits and follow-up visits to include neurocognitive testing, VO2 max testing (graded exercise test), blood draws, and retinal scans. Potential subjects must pass an exercise stress test with 12-lead ECG, and training sessions (exercise protocol). Standardized neurocognitive tests assessing functions such as memory and attention will be administered and retinal scans will be conducted. The at-home exercise intervention will be supervised via the Polar beat/flow applications by study personnel. Subjects will engage in cardiovascular exercise with heart rate monitoring on 4 days per week for a total of 10 weeks.
  Interventions: Other: High Intensity Interval Training (HIIT) Exercise

INTERVENTIONS:
Other: High Intensity Interval Training (HIIT) Exercise — Participants will exercise 4 days/week for 10 weeks using the High Intensity Interval Training (HIIT) protocol. Sessions can be conducted at home or at a gym with access to a cycle ergometer. Participants will undergo 2 supervised training sessions to learn the HIIT protocol. To record heart rate, session duration, and time at each exercise intensity, participants will be provided with an H10 Polar TM heart rate chest strap monitor and a Polar Beat/Polar Flow account. Participants will download the Polar Beat/Flow smart phone application to record exercise sessions and allow the researcher to conduct remote data monitoring. Research staff will contact participants twice per week to provide feedback.

SUMMARY:
The investigator aims to assess the extent to which a brief exercise intervention improves systemic growth factor concentrations, reverses loss of systemic vascular networks and hypertension, and by extension, improves neurocognition. To test the investigator's hypothesis that increased cardiovascular fitness will correlate with improved vascular density, the investigator proposes the innovative use of retinal density scans.

ELIGIBILITY:
Inclusion Criteria:

* adults between 55-75 years of age
* essential hypertension (as determined by referring physicians)
* engages in less than 150 minutes of moderate intensity exercise/week (as determined by CHAMPS Questionnaire)
* physically able to exercise
* access to an upright cycle ergometer at home or via gym access
* access to smart device (iOS or Android phone or tablet with ability to install and use Polar Beat and Polar FlowTM applications).

Exclusion Criteria:

* diagnosis of dementia
* resting systolic blood pressure <120, or >180 mm Hg
* disease or condition that would preclude exercise
* untreated depression or anxiety disorders
* severe respiratory disease
* disease of the eye
* refractive error > 6 diopters or +6 diopters (as assessed by 1st retinal scan).

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Changes in graded exercise stress test | 16 weeks
  This test will measure participants' maximal oxygen utilization and will be done once before and once after exercise intervention. The investigator will use a graded exercise test on a stationary cycle. The test will continue to maximum, and expired gases will be collected (via a spirometer) throughout the test to monitor oxygen consumption and carbon dioxide expiration. The investigator defines maximum or test termination as either voluntary exhaustion by the participant, or by two of three physiologic criteria: 1) heart rate = 220 minus age; 2) respiratory exchange ratio > 1.15; 3) Stabilization of oxygen consumption with increasing workload. The participant's effort is monitored at each test stage via the standard 6-20 rating of a perceived exertion scale. Lactate levels will also be collected by finger prick to help determine maximum.
Retinal microvascular density changes | 16 weeks
  Standardized Optical Coherence Tomography Angiography (OCT-A) scans will occur twice before and once after exercise intervention to measure retinal microvascular density changes. A fractal analysis will be used to uniquely analyze the retinal microvascular network so that global changes of the vascular system can be quantified.
Cognitive changes | 16 weeks
  Standardized neuropsychological tests will be completed twice before and once after exercise intervention. These are designed to assess global functions of processing speed, memory, attention, and executive function, which have been shown to be sensitive to diffuse effects of cardiogenic, cerebral hypoperfusion. All tests have published, aged-adjusted norms. Specific tests include: Trail making A & B, Digit Span; Rey Complex Figure (RCFT); Digit Symbol; Controlled Oral Word Association (verbal fluency); Hopkins Verbal Learning Test (HVLT); Boston Naming Test; Center for Epidemiologic Studies-Depression Scale (CES-D), and the Brief Visual Memory Test (BVMT). At each time point, the Z scores for all measures will be aggregated and divided by 9 to arrive at the total cognitive Z-score. In addition, we will calculate composite scores for separate cognitive domains using the same approach and compare each time point to measure total cognitive changes.
Serum growth factor changes | 16 weeks
  Approximately 2 teaspoons (10 mL) of venous blood draw will occur twice before and once after exercise intervention to measure serum growth factor changes.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Lazar, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No